CLINICAL TRIAL: NCT06674369
Title: Timlioğlu İper H.S1, Sahli.E2, İdil Ş.A3,Önal.R.E4 1 PhD.MD Opht.İstanbul Okan University ,ophthalmology and Opticianry ,ORCİD:0000-0003-2112-0602 2 PhD.MD Opht. Ankara University Faculty of Medicine, Low Vision Rehabilitation and Research Center, Department of Ophthalmology, Ankara, Turkey ORCİD:0000-0002-1355-7284 3 MD Opht. Professor. Ankara University Faculty of Medicine, Low Vision Rehabilitation and Research Center, Department of Ophtha
Brief Title: Ongoing Effect of Expansion Prisms Following the Discontinuation of Use on Visual Field Enlargement and Retrograde Ganglion Cell Degeneration in Homonymous Hemianopia Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Okan University (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, Hatice Semrin Timlioglu İper, Assistant Professor, Okan University
Other Study IDs: 24.08.2022/20
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-09

CONDITIONS: Homonymous Hemianopsia
Keywords: Homonium hemianopsia; Retrograde ganglion cell degeneration; Neuroplastisity,; Vision therapy,; Peli Prism
MeSH Terms: conditions — Hemianopsia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 15 patients between the ages of 22-70 (m=52.0 year) with homonymous hemianopsia: Homonymous hemianopia (HH) patients due to long-standing post-chiasmatic lesions between 2017 and 2020 were included in the study . To eliminate spontaneous neuronal recovery only the patients with hemianopia, diagnosed at least six months before the initial examination and who had undergone full clinical MRI evaluation were included. Initially all patients were applied peripheral field expander 40 D horizontal Peli prisms. In the initial and follow-up examinations, in addition to neurological history, a complete ophthalmologic examination was performed, followed by computerized visual field examination using Estermann binocular field program and Swedish Interactive treshold algorithm program (SITA 30-2) (Zeiss Humphrey3-850). Ganglion cell layer thickness was measured by OCT (Zeiss Cirrus HD Oct) and compared with the normal retinal image.
  Interventions: Device: Peli prism for hemianopia

INTERVENTIONS:
Device: Peli prism for hemianopia — Peli prism uses high-powered prisms (40 Dioptre) that expand a hemianopic patient's awareness of their blind side. This awareness enables patients to better detect obstacles and navigate around them. Effect of the prism considered as temporary We investigated whether the effect persists after the prism is removed.To understand the persistence of the effect, we examined the changes in the visual field with CVF (Computerized visual field examination)before the prism was applied, with the prism and 1 week after the prism was removed.
  Other Names: Computerised visual filed examination; Optic coherence tomography

SUMMARY:
The goal of this observational study is to learn about the long-term effects of Pelli prism in Hemianopia patients who take Prisms for awareness of the area they cannot see.

The main question it aims to answer is:

Does the field enlargement observed with the prism continues after the prism is removed? Participants already using Peli prisms as part of their regular medical care for Hemianopia, in the upcoming routine controls their field of vision enlargements will be examined.

DETAILED DESCRIPTION:
Hemianopia is a disability-causing condition that usually affects young to middle-aged people and reduces quality of life.Prism applications are one of the rehabilitation methods used to improve the quality of life of these people and ensure their participation in daily life. The Peli prism is the most commonly used prism type. The effect of prism applications is thought to be temporary.The main idea of our study is that Prisms can create longlasting effects by affecting neuroplasticity.

ELIGIBILITY:
Inclusion Criteria:

Homonim Hemianopsia patient age between 18-55 years H.Hemianopia, diagnosed at least six months before the initial examination Neurological condition is suitable for daily activities

Exclusion Criteria:

- Failure to meet age criteria Hemianopia developed more recently than 6 months ago Having to use medications that affect his/her balance and daily activity

Ages: 18 Months to 55 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hemianopia patients admitted to the ophthalmology clinic of Okan University Hospital and the ophthalmology clinic of Ankara University Faculty of Medicine were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Computerised visual field changes | From enrollment to the end of prism use at 6 months
  Changes in Visual field index(VFİ) and mean devation(MD) in dB. Higher values in VFI and MD mean an improvement in visual field

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Sefay İdil, Professor, Study Director — Ankara Üniversity
Locations (1):
- Okan University Hospital Ophthalmology clinic, Istanbul, Tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2.12.2024
Access Criteria: Open access for academics

REFERENCES:
- [Background] Garric C, Sebaa A, Caetta F, Perez C, Savatovsky J, Sergent C, Chokron S. Dissociation between objective and subjective perceptual experiences in a population of hemianopic patients: A new form of blindsight? Cortex. 2019 Aug;117:299-310. doi: 10.1016/j.cortex.2019.05.006. Epub 2019 May 18. PMID 31181393
- See also: The risk of pedestrian collisions with peripheral visual field loss. Journal of vision, 16(15), 5-5 — https://doi.org/10.1167/16.15.5